CLINICAL TRIAL: NCT01622712
Title: Evaluation of Mesh Integration and Mesh Contraction After Open Preperitoneal Inguinal Hernia Repair Using a Memory Ring Containing Device.
Acronym: REBOUND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Medri (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011/823
Record Dates: First submitted 2012-06-15; First posted 2012-06-19 (Estimated); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Unilateral Inguinal Hernia
Keywords: inguinal hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Unilateral inguinal hernia (Experimental): A Nitinol containing large pore polypropylene mesh will be placed in patients with unilateral inguinal hernia.
  Interventions: Device: Rebound HRD Mesh

INTERVENTIONS:
Device: Rebound HRD Mesh — Patients with unilateral inguinal hernia receive a nitinol containing large pore polypropylene mesh.

SUMMARY:
The aim of this study is to evaluate whether preperitoneal mesh placement using a nitinol containing large pore polypropylene mesh (REBOUND HRD™) offers a satisfying patient recovery, quick reconvalescence and adequate tissue integration with acceptable mesh contraction in a multicenter (Belgian) prospective trial.

Patients treated by open preperitoneal mesh repair for an unilateral inguinal hernia according the current surgical practice in the participating centers will be observed during one year post-surgery, after which they will have a CT scan of the surgical area in the groin to evaluate the mesh changes regarding shrinkage and migration.

ELIGIBILITY:
Inclusion Criteria:

* elective repair for a primary unilateral inguinal hernia OR
* elective repair for a recurrent unilateral inguinal hernia after non-mesh repair

Exclusion Criteria:

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2014-09-02 (Actual); Study Completion 2014-09-02 (Actual)

PRIMARY OUTCOMES:
Calculation and measurement of shrinkage (%) of mesh surface after surgical mesh implantation. | 12 months post-surgery
  A CT scan is performed.

SECONDARY OUTCOMES:
Pain assessment. | after 1 year
Discomfort assessment. | after 1 year
Use of oral analgetics. | after 1 year
Wound morbidity. | after 4 weeks
Recurrence of hernia. | after 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Berrevoet, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (2):
- Belgium (2):
  - ASZ Aalst, Aalst
  - Ghent University Hospital, Ghent

REFERENCES:
- See also: Related Info — http://www.uzgent.be